CLINICAL TRIAL: NCT06846203
Title: Comparison of Core Stabilization and Neuromuscular Facilitation Exercises for Lowback Pain Prevention Among Health Care Professionals
Brief Title: Comparison of Core Stabilization and Neuromuscular Facilitation Exercises for Lowback Pain Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Riphah Mehreen Raza
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Postural Low Back Pain
Keywords: Dynamic sit up test; Low Back Pain; Functional Movement Screen; PNF stretching exercises
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stabilization exercises (Experimental): This group will be subjected to following core stabilization exercises which include Sit-up-1, Sit-up-2, Back extention-1,Back extention-2 , Front plank,Back bridge ,Quadruped and Side bridge.
  Interventions: Other: Core stabilization Exercise Group
- Neuromuscular Fascilitation exercises (Experimental): This group will be subjected to neuromuscular facilitation exercises which includes McGill curl up,Bird dog stretch, Side bridge or mermaid side bridge with bent knees, Single leg stretching ,Shoulder bridge,"Tai chi Warrior" stance ,Cat - cow - downward facing dog, Hip circumduction, hamstring stretching and starting position.
  Interventions: Other: Neuromuscular Fascilitation Exercise Group

INTERVENTIONS:
Other: Core stabilization Exercise Group — This group will be subjected to following core stabilization exercises:
  1: Sit-up-1, 2: Sit-up-2, 3: Back extention-1, 4: Back extention-2 , 5: Front plank, 6: Back bridge , 7: Quadruped , 8:Side bridge A combination of activities will be administered and alterations will be made every session.
  Session will be held 3 times per week for 8 consecutive weeks.
  Arms: core stabilization exercises
Other: Neuromuscular Fascilitation Exercise Group — This group will be subjected to neuromuscular facilitation exercises :
  Week 1: McGill curl up, Week 2: Bird dog stretch, Week 3: Side bridge or mermaid side bridge with bent knees, Week 4: Single leg stretching, Week 5: Shoulder bridge Week 6: "Tai chi Warrior" stance, Week 7 & 8: Cat - cow - downward facing dog, Hip circumduction, hamstring stretching, starting position Session will be held 3 times per week for 8 consecutive weeks
  Arms: Neuromuscular Fascilitation exercises

SUMMARY:
Low back pain (LBP) is a leading cause of disability worldwide, particularly affecting individuals in occupations that demand prolonged sitting or standing, such as healthcare professionals. The nature of their work often involves sustained postures, physical exertion, and repetitive movements, which compromise core muscle function and neuromuscular control, increasing the risk of spinal dysfunction and pain. Core stabilization exercises have been widely recognized for their role in improving trunk strength, enhancing postural alignment, and reducing spinal loading, thereby preventing LBP. Similarly, neuromuscular facilitation exercises aim to optimize muscle activation patterns, improve coordination, and restore functional movement, making them a promising strategy for LBP prevention. Despite the individual benefits of these approaches, there is a paucity of comparative research investigating their relative effectiveness in the prevention of LBP, particularly in populations with demanding physical and postural requirements, such as healthcare professionals.

This study seeks to fill this gap by comparing the effects of core stabilization exercises and neuromuscular facilitation exercises on LBP prevention among healthcare professionals.The findings will provide evidence-based guidance for designing targeted interventions, ultimately promoting musculoskeletal health and enhancing the occupational well-being of this vulnerable group.

DETAILED DESCRIPTION:
Healthcare professionals perform daily activities that can lead to musculoskeletal disorders among them the lower back, neck, shoulder and hand/wrist are the most exposed areas.Healthcare professionals frequently engage in activities that require lifting, bending, and prolonged standing or sitting, which can place significant stress on their lower back .Low back pain is prevalent among healthcare workers, with studies indicating that over 57% of professionals experience it at some point in their careers Contributing factors include prolonged standing, frequent bending and twisting, and the physical demands of nursing and medical roles .The prevalence is notably higher among healthcare professionals, highlighting the need for targeted prevention strategies.

Researches have been done in order to devise strategies for the reduction of low back pain. Core stabilization and Neuromuscular Facilitation exercises are among them. Research shows that core stability training can alleviate symptoms of nonspecific low back pain (NSLBP) in nurses by improving muscle endurance and balance between the multifidus muscles on both sides of the spine Engaging in regular physical activity, including stretching exercises, has been shown to reduce LBP symptoms and improve overall physical health. For instance, a study found that a structured stretching program significantly reduced pain levels among healthcare workers .Core strengthening exercises, which include the muscles of the abdomen, pelvis, and lower back, are crucial for maintaining spinal stability and preventing LBP. likewise propioceptive neuromuscular fascilitation exercises have been shown to improve trunk muscle endurance and strength, which are critical for supporting the lumbar spine. Studies found that participants engaging in Propioceptive neuromuscular fascilitation demonstrated substantial gains in trunk stability and mobility, essential factors in preventing future episodes of back pain .

Evidence suggests that the benefits of Neuromuscular Fascilitation may extend beyond immediate pain relief, contributing to long-term improvements in muscle activity and overall spinal health. A study highlighted that PNF can lead to sustained reductions in pain and increases in functional capacity over time. When compared with traditional core strengthening exercises or conventional physical therapy, Neuromuscular Fascilitation has shown superior outcomes in terms of both pain reduction and functional improvement.This positions Neuromuscular Fascilitation as a potentially more effective intervention for healthcare professionals who are at risk for developing LBP.An RCT was conducted by waseem et al in 2017 inorder to compare core stabilization exercises with conventional physical therapy.They concluded that clinical and therapeutic effects of core stabilization exercise program over the period of six weeks are more effective in terms of reduction in pain, compared to routine physical therapy exercise for similar duration. Pattanasin et al compared core stabilization exercises with Neuromuscular Fascilitation and reported that four-week Core stabilization and neuromuscular fascilitation training provided short-term and long-term effects on pain-related outcomes, along with increased deep trunk muscle activity in Chronic low back patients.Su et al in a study conducted in 2021 reported that Despite both core stabilization and strengthening exercises reducing pain, core stabilization exercise is superior to strengthening exercise. It is effective in improving proprioception, balance, and percentage change of muscle thickness of TrA and LM, and reducing functional disability and ear of movement in patients with subacute Non specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Professionals including nurses, dentist, surgeons, physiotherapists etc.
* 20-45 years.
* Both genders.
* Individuals with no back pain history from previous 3 months.
* Individuals having Biering sorensen test score less than 176 seconds.

Exclusion Criteria:

* Individuals who had experienced low back pain in previous 3 months.
* Diagnosed musculoskeletal and neuromuscular problems.
* Diagnosed cardiovascular or pulmonary problems.
* Any Fractures and spine surgery.
* Individuals who are already a part of any interventional research program.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Dynamic Sit Up Test. | Baseline to 8th week
  The Dynamic Situp Test evaluates the endurance of the abdominal muscles and consists of consecutive performance of 3 increasingly difficult kinds of sit-up, 5 repetitions each. The examinee lies face-up on the floor with the knees bent at 90 degrees and the feet flat on the floor, held down by an examiner. The examinee then attempts to perform 15 situps in the following sequence. There should be no rest period or pause between the different types of sit-up:
  5 situps each with the hands sliding along the thighs,while keeping the forearms crossed over the chest and with the fingertips maintaining contact with the back of the earlobes.
  The score is the total number of situps performed (max = 15) A Cronbach's alpha reliability analysis of the entire sample revealed a high degree of interrater reliability for the sit-up test. (α = .925)
Biering sorenson Test. | Baseline to 8th week
  The Biering-Sørensen test is commonly used to assess endurance of the paraspinal musculature using two metrics: test duration (the time that an individual maintains the Sørensen test position), and rate of muscle fatigue it is reported to predict low back pain within the next year in males. The test consists in measuring the amount of time a person can hold the unsupported upper body in a horizontal prone position with the lower body fixed to the examining table For the Sørensen tests, participants lay on a Roman chair with their lower limbs stabilized and their head, arms, and trunk unsupported. Participants were instructed to maintain a horizontal body position for as long as possible. The end of the test occurred when the participant could no longer maintain the horizontal test position or when the participant felt unable to continue the test. A low Biering-Sorensen score has been found to predict who will have nonspecific low back pain.
Functional movement Screen. | Baseline to 8th week
  The Functional Movement Screen (FMS) is a screening system that attempts allow the professional to assess the fundamental movement patterns of an individual. Its seven components are: Deep Squat, Hurdle Step, and In-Line Lunge, Shoulder Mobility, the Active Straight Leg Raise, the Trunk Stability Push-up, and Rotary Stability The maximum possible score on the FMS is 21, which is achieved by scoring a perfect 3 on all seven tests. Conversely, a score below 14 suggests a higher risk for injury due to poor body mechanics.The FMS demonstrates good to excellent interrater reliability, with intraclass correlation coefficients (ICCs) reported between 0.76 and 0.98 across various studies.The FMS has shown predictive validity for injury risk, particularly with a composite score of ≤14, which indicates a significantly higher likelihood of sustaining injuries .

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International Hospital, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No